CLINICAL TRIAL: NCT01587079
Title: A Randomized, Double Blind, (Test Products), Chronic Dosing (7 Days), Four Period, Eight Treatment , Incomplete Block, Cross Over, Multi Center Study to Assess Efficacy and Safety of Five Doses of PT003, One Dose of PT001 and One Dose of PT005 in Patients With Moderate to Severe COPD, Compared With Spiriva® Handihaler® (Tiotropium Bromide 18 µg, Open Label) as Active Control
Brief Title: Glycopyrrolate/Formoterol Fumarate MDI Compared With Spiriva® as An Active Control in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT003005
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Results first posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- PT003 (Dose 1) (Experimental): PT003 MDI Dose 1
  Interventions: Drug: PT003
- PT003 (Dose 2) (Experimental): PT003 MDI Dose 2
  Interventions: Drug: PT003
- PT003 (Dose 3) (Experimental): PT003 MDI Dose 3
  Interventions: Drug: PT003
- PT003 (Dose 4) (Experimental): PT003 MDI Dose 4
  Interventions: Drug: PT003
- PT003 (Dose 5) (Experimental): PT003 MDI Dose 5
  Interventions: Drug: PT003
- PT001 (Experimental): PT001 MDI
  Interventions: Drug: PT001
- PT005 (Experimental): PT005 MDI
  Interventions: Drug: PT005
- Spiriva® Handihaler® (Active Comparator): Tiotropium Bromide
  Interventions: Drug: Tiotropium inhalation powder

INTERVENTIONS:
Drug: PT003 — PT003 MDI administered as two puffs BID for 7 days
  Arms: PT003 (Dose 1); PT003 (Dose 2); PT003 (Dose 3); PT003 (Dose 4); PT003 (Dose 5)
Drug: PT001 — PT001 MDI administered as two puffs BID for 7 days
  Arms: PT001
Drug: PT005 — PT005 MDI administered as two puffs BID for 7 days
  Arms: PT005
Drug: Tiotropium inhalation powder — Taken as 1 capsule containing 18 µg of Tiotropium via the Handihaler DPI for 7 days
  Arms: Spiriva® Handihaler®

SUMMARY:
The primary objective of this study is to assess the efficacy of Glycopyrrolate/Formoterol Fumarate MDI relative to individual components (GP MDI and FF MDI) in subjects with moderate to severe COPD

ELIGIBILITY:
Key Inclusion Criteria:

* Signed written informed consent
* 40 - 80 years of age
* Clinical history of COPD with airflow limitation that is not fully reversible
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test and acceptable contraceptive methods
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* A measured post-bronchodilator FEV1/FVC ratio of < or = 0.70
* A measured post-bronchodilator FEV1 > or = 750ml or 30% predicted and < or = 80% of predicted normal values
* Able to change COPD treatment as required by protocol

Key Exclusion Criteria:

* Women who are pregnant or lactating
* Primary diagnosis of asthma
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Active pulmonary diseases
* Prior lung volume reduction surgery
* Abnormal chest X-ray not due to the presence of COPD
* Hospitalized due to poorly controlled COPD within 3 months of Screening
* Clinically significant medical conditions that preclude participation in the study (e.g. clinically significant abnormal ECG, uncontrolled hypertension, glaucoma, symptomatic prostatic hypertrophy)
* Cancer that has not been in complete remission for at least 5 years
* Treatment with investigational study drug or participation in another clinical trial or study within the last 30 days or 5 half lives

Other inclusion/exclusion criteria as defined in the protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Director — Pearl Therapeutics, Inc.
Locations (17):
- United States (17):
  - Pearl Investigative Site, Glendale, Arizona
  - Pearl Investigative Site, Rancho Mirage, California
  - Pearl Investigative Site, Waterbury, Connecticut
  - Pearl Investigative Site, Clearwater, Florida
  - Pearl Investigative Site, Pensacola, Florida
  - Pearl Investigative Site, Winter Park, Florida
  - Pearl Investigative Site, Lafayette, Louisiana
  - Pearl Investigative Site, North Dartmouth, Massachusetts
  - Pearl Investigative Site, Fridley, Minnesota
  - Pearl Investigative Site, St Louis, Missouri
  - Pearl Investigative Site, Summit, New Jersey
  - Pearl Investigative Site, Cincinnati, Ohio
  - Pearl Investigative Site, Medford, Oregon
  - Pearl Investigative Site, Rock Hill, South Carolina
  - Pearl Investigative Site, Spartanburg, South Carolina
  - Pearl Investigative Site, San Antonio, Texas
  - Pearl Investigative Site, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 sites in the US from May 2012 until September 2012. The entire study was scheduled to take a maximum of 19 weeks for each individual subject.
Pre-assignment Details: Study was a chronic dosing (7 days), 4-period, 8-treatment, Incomplete Block, Cross-Over.
Period: Overall Study
Arm/Group | All Subjects
Started | 159
Completed | 120
Not Completed | 39
Not completed — Protocol-specified criteria | 9
Not completed — Protocol Violation | 5
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 14

BASELINE CHARACTERISTICS:
Population: ITT/Safety Population
Arm/Group | All Subjects Screened
Number analyzed (Participants) | 159
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age, years | 62.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 (47.8)
  Male | 83 (52.2)

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC 0-12 on Day 7
Description: FEV1 AUC 0-12
Time Frame: Day 7
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- GP MDI 18 μg (PT001): 18 μg
- GFF MDI 18/9.6 μg (PT003): 18/9.6 μg
- GFF/MDI 9/9.6 μg: 9/9.6 μg
- GFF MDI BID 4.6/9.6 μg: 4.6/9.6 μg
- GFF MDI 2.4/9.6 μg (PT003): 2.4/9.6 μg
- GFF MDI 1.2/9.6 μg (PT003): 1.2/9.6 μg
- FF MDI 9.6 μg: 9.6 μg
- Spiriva 18 μg QD: 18 μg QD
Arm/Group | GP MDI 18 μg (PT001) | GFF MDI 18/9.6 μg (PT003) | GFF/MDI 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI 2.4/9.6 μg (PT003) | GFF MDI 1.2/9.6 μg (PT003) | FF MDI 9.6 μg | Spiriva 18 μg QD
Number analyzed (Participants) | 57 | 59 | 52 | 57 | 57 | 60 | 57 | 60
Liters | 1.452 [1.415 to 1.489] | 1.591 [1.554 to 1.628] | 1.547 [1.509 to 1.585] | 1.539 [1.502 to 1.575] | 1.538 [1.502 to 1.575] | 1.508 [1.472 to 1.545] | 1.467 [1.430 to 1.505] | 1.489 [1.453 to 1.525]

2. Secondary Outcome: Peak Change From Baseline in FEV1 on Treatment Day 1
Description: Peak change from Baseline in FEV1 on Treatment
Time Frame: Day 1
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Milliliters
Groups:
- GP MDI BID 18 μg: BID 18 μg
- GFF MDI BID 18/9.6 μg: BID 18/9.6 μg
- GFF/MDI BID 9/9.6 μg: BID 9/9.6 μg
- GFF MDI BID 2.4/9.6 μg: BID 2.4/9.6 μg
- GFF MDI BID 1.2/9.6 μg: BID 1.2/9.6 μg
- FF MDI BID 9.6 μg: BID 9.6 μg
Arm/Group | GP MDI BID 18 μg | GFF MDI BID 18/9.6 μg | GFF/MDI BID 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI BID 2.4/9.6 μg | GFF MDI BID 1.2/9.6 μg | FF MDI BID 9.6 μg | Spiriva 18 μg QD
Number analyzed (Participants) | 59 | 63 | 56 | 60 | 60 | 64 | 59 | 63
Milliliters | 209 [172 to 246] | 339 [302 to 376] | 329 [292 to 367] | 348 [311 to 386] | 333 [296 to 370] | 312 [275 to 349] | 317 [280 to 355] | 238 [201 to 274]

3. Secondary Outcome: Time to Onset of Action (>10% Improvement in FEV1) on Day 1
Description: Time to onset of action (>10% improvement in FEV1)
Time Frame: Day 1
Population: MITT
Measure: Number; unit: Percentage
Arm/Group | GP MDI BID 18 μg | GFF MDI BID 18/9.6 μg | GFF/MDI BID 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI BID 2.4/9.6 μg | GFF MDI BID 1.2/9.6 μg | FF MDI BID 9.6 μg | Spiriva 18 μg QD
Number analyzed (Participants) | 60 | 62 | 55 | 58 | 60 | 64 | 60 | 62
Percentage
  15 minutes | 27 | 65 | 51 | 62 | 65 | 66 | 60 | 37
  30 minutes | 8 | 18 | 13 | 10 | 10 | 9 | 3 | 21
  1 hour | 15 | 6 | 11 | 12 | 12 | 5 | 12 | 11
  2 hours | 10 | 5 | 7 | 5 | 2 | 9 | 3 | 5
  No onset within 2 hours | 40 | 6 | 18 | 10 | 12 | 11 | 22 | 26

4. Secondary Outcome: Proportion of Subjects Achieving >=12% Improvement in FEV1 on Day 1
Description: Proportion of subjects achieving >=12% improvement in FEV1
Time Frame: Day 1
Population: MITT
Measure: Number; unit: Percentage
Arm/Group | GP MDI BID 18 μg | GFF MDI BID 18/9.6 μg | GFF/MDI BID 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI BID 2.4/9.6 μg | GFF MDI BID 1.2/9.6 μg | FF MDI BID 9.6 μg | GP MDI 18 μg (PT001)
Number analyzed (Participants) | 60 | 63 | 55 | 59 | 61 | 65 | 61 | 63
Percentage | 56 | 93 | 85 | 84 | 86 | 83 | 80 | 72

5. Secondary Outcome: Peak Change From Baseline in Inspiratory Capacity on Day 1
Description: Peak change from baseline in Inspiratory Capacity
Time Frame: Day 1
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Milliliters
Arm/Group | GP MDI BID 18 μg | GFF MDI BID 18/9.6 μg | GFF/MDI BID 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI BID 2.4/9.6 μg | GFF MDI BID 1.2/9.6 μg | FF MDI BID 9.6 μg | Spiriva 18 μg QD
Number analyzed (Participants) | 60 | 63 | 56 | 61 | 61 | 65 | 62 | 63
Milliliters | 204 [131 to 278] | 393 [320 to 467] | 320 [244 to 397] | 387 [313 to 461] | 347 [274 to 421] | 348 [276 to 420] | 335 [261 to 409] | 233 [160 to 305]

6. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 on Day 7
Description: Change from baseline in morning pre-dose trough FEV1
Time Frame: Day 7
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Milliliters
Arm/Group | GP MDI BID 18 μg | GFF MDI BID 18/9.6 μg | GFF/MDI BID 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI BID 2.4/9.6 μg | GFF MDI BID 1.2/9.6 μg | FF MDI BID 9.6 μg | Spiriva 18 μg QD
Number analyzed (Participants) | 60 | 62 | 56 | 61 | 60 | 65 | 60 | 63
Milliliters | 120 [87 to 152] | 183 [151 to 216] | 150 [117 to 184] | 154 [121 to 186] | 163 [130 to 195] | 130 [98 to 162] | 104 [71 to 137] | 122 [90 to 155]

7. Secondary Outcome: Peak Change From Baseline in FEV1 on Day 7
Description: Peak change from baseline in FEV1 Day 7
Time Frame: Day 7
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Millliters
Arm/Group | GP MDI BID 18 μg | GFF MDI BID 18/9.6 μg | GFF/MDI BID 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI BID 2.4/9.6 μg | GFF MDI BID 1.2/9.6 μg | FF MDI BID 9.6 μg | Spiriva 18 μg QD
Number analyzed (Participants) | 60 | 63 | 55 | 60 | 61 | 64 | 60 | 63
Millliters | 300 [257 to 342] | 444 [402 to 487] | 414 [370 to 458] | 403 [361 to 446] | 388 [345 to 430] | 363 [321 to 404] | 332 [289 to 375] | 309 [267 to 351]

8. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough IC on Day 7
Description: Change from baseline in morning pre-dose trough IC
Time Frame: Day 7
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Millliters
Arm/Group | GP MDI BID 18 μg | GFF MDI BID 18/9.6 μg | GFF/MDI BID 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI BID 2.4/9.6 μg | GFF MDI BID 1.2/9.6 μg | FF MDI BID 9.6 μg | Spiriva 18 μg QD
Number analyzed (Participants) | 60 | 63 | 56 | 61 | 61 | 63 | 62 | 63
Millliters | 109 [46 to 171] | 185 [123 to 246] | 183 [119 to 247] | 215 [153 to 278] | 203 [141 to 265] | 151 [89 to 212] | 129 [67 to 191] | 106 [45 to 168]

9. Secondary Outcome: Peak Change From Baseline IC on Day 7
Description: Peak change from baseline IC
Time Frame: Day 7
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Millliters
Arm/Group | GP MDI BID 18 μg | GFF MDI BID 18/9.6 μg | GFF/MDI BID 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI BID 2.4/9.6 μg | GFF MDI BID 1.2/9.6 μg | FF MDI BID 9.6 μg | Spiriva 18 μg QD
Number analyzed (Participants) | 60 | 63 | 56 | 61 | 61 | 65 | 62 | 63
Millliters | 223 [149 to 297] | 430 [357 to 503] | 441 [366 to 516] | 409 [335 to 484] | 368 [294 to 441] | 371 [298 to 444] | 377 [303 to 452] | 241 [168 to 314]

10. Secondary Outcome: Change From Baseline at Evening 12-hour Post-dose Trough FEV1 on Day 7
Description: Change from baseline at evening 12-hour post-dose trough FEV1
Time Frame: Day 7
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Millliters
Arm/Group | GP MDI BID 18 μg | GFF MDI BID 18/9.6 μg | GFF/MDI BID 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI BID 2.4/9.6 μg | GFF MDI BID 1.2/9.6 μg | FF MDI BID 9.6 μg | Spiriva 18 μg QD
Number analyzed (Participants) | 57 | 61 | 53 | 59 | 57 | 61 | 59 | 61
Millliters | 99 [53 to 145] | 196 [151 to 241] | 162 [115 to 209] | 118 [73 to 163] | 133 [87 to 179] | 110 [65 to 155] | 73 [28 to 119] | 130 [85 to 174]

11. Secondary Outcome: Change From Baseline in Mean Morning Pre-dose Daily Peak Flow Readings on Day 7
Description: Change from baseline in mean morning pre-dose daily peak flow readings
Time Frame: Day 7
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Groups:
- GP MDI 18 μg BID: 18 μg BID
- GFF MDI 18/9.6 μg BID: 18/9.6 μg BID
- GFF/MDI 9/9.6 μg BID: 9/9.6 μg BID
- GFF MDI 2.4/9.6 μg BID: 2.4/9.6 μg BID
- GFF MDI 1.2/9.6 μg BID: 1.2/9.6 μg BID
- FF MDI 9.6 μg BID: 9.6 μg BID
Arm/Group | GP MDI 18 μg BID | GFF MDI 18/9.6 μg BID | GFF/MDI 9/9.6 μg BID | GFF MDI BID 4.6/9.6 μg | GFF MDI 2.4/9.6 μg BID | GFF MDI 1.2/9.6 μg BID | FF MDI 9.6 μg BID | Spiriva 18 μg QD
Number analyzed (Participants) | 59 | 63 | 56 | 61 | 61 | 64 | 62 | 62
L/min | 7.6 [0.5 to 14.8] | 25.2 [18.1 to 32.4] | 16.6 [9.4 to 23.9] | 12.4 [5.2 to 19.5] | 18.0 [10.9 to 25.1] | 13.8 [6.7 to 20.8] | 8.6 [1.5 to 15.7] | 11.6 [4.5 to 18.7]

12. Secondary Outcome: Change From Baseline in Mean Morning Post-dose Daily Peak Flow Readings on Day 7
Description: Change from baseline in mean morning post-dose daily peak flow readings on
Time Frame: Day 7
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | GP MDI 18 μg BID | GFF MDI BID 18/9.6 μg | GFF/MDI BID 9/9.6 μg | GFF MDI BID 4.6/9.6 μg | GFF MDI BID 2.4/9.6 μg | GFF MDI 1.2/9.6 μg BID | FF MDI 9.6 μg BID | Spiriva 18 μg QD
Number analyzed (Participants) | 59 | 62 | 56 | 61 | 61 | 64 | 62 | 62
L/min | 31.0 [23.0 to 39.0] | 58.8 [50.9 to 66.7] | 55.0 [46.9 to 63.1] | 46.7 [38.8 to 54.6] | 52.1 [44.1 to 60.0] | 49.6 [41.7 to 57.4] | 43.2 [35.3 to 51.1] | 37.9 [30.0 to 45.8]

13. Secondary Outcome: Change From Baseline in Mean Evening Pre-dose Daily Peak Flow Readings on Day 7
Description: Change from baseline in mean evening pre-dose daily peak flow readings (BID treatments only)
Time Frame: Day 7
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Groups:
- GFF MDI 4.6/9.6 μg BID: 4.6/9.6 μg BID
- Spiriva18 μg QD: 18 μg QD
Arm/Group | GP MDI 18 μg BID | GFF MDI 18/9.6 μg BID | GFF/MDI 9/9.6 μg BID | GFF MDI 4.6/9.6 μg BID | GFF MDI 2.4/9.6 μg BID | GFF MDI 1.2/9.6 μg BID | FF MDI 9.6 μg BID | Spiriva18 μg QD
Number analyzed (Participants) | 57 | 59 | 56 | 58 | 60 | 63 | 62 | 0
L/min | 11.7 [4.6 to 18.7] | 32.5 [25.4 to 39.5] | 25.0 [18.0 to 32.1] | 19.0 [12.0 to 26.0] | 25.6 [18.7 to 32.5] | 19.9 [13.0 to 26.8] | 16.5 [9.6 to 23.4] |

14. Secondary Outcome: Change From Baseline in Mean Evening Post-dose Daily Peak Flow Readings on Day 7
Description: Change from baseline in mean evening post-dose daily peak flow readings (12 Hours post-dose for Spiriva)
Time Frame: Day 7
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Groups:
- GFF MDI BID 4.6/9.6 μg BID: 4.6/9.6 μg BID
Arm/Group | GP MDI 18 μg BID | GFF MDI 18/9.6 μg BID | GFF/MDI 9/9.6 μg BID | GFF MDI BID 4.6/9.6 μg BID | GFF MDI 2.4/9.6 μg BID | GFF MDI 1.2/9.6 μg BID | FF MDI 9.6 μg BID | Spiriva 18 μg QD
Number analyzed (Participants) | 57 | 57 | 56 | 58 | 60 | 63 | 62 | 60
L/min | 35.0 [26.8 to 43.2] | 61.5 [53.1 to 69.8] | 56.1 [47.8 to 64.3] | 51.5 [43.3 to 59.7] | 53.7 [45.6 to 61.7] | 53.8 [45.8 to 61.8] | 48.3 [40.3 to 56.4] | 30.3 [22.2 to 38.4]

ADVERSE EVENTS:
Time Frame: SAEs and AEs were collected throughout study participation and up to 14 days following the last dose of study drug.
Description: Safety Population - All subjects who were randomized, received at least 1 dose of a study treatment, and had a post-baseline safety assessment for that treatment.
Groups:
- GFF MDI 9/9.6 μg (PT003): 9/9.6 μg
- GFF MDI 4.6/9.6 μg (PT003): 4.6/9.6 μg
- FF MDI 9.6 μg (PT005): 9.6 μg
- Spiriva: 18 μg
Arm/Group | GP MDI 18 μg (PT001) | GFF MDI 18/9.6 μg (PT003) | GFF MDI 9/9.6 μg (PT003) | GFF MDI 4.6/9.6 μg (PT003) | GFF MDI 2.4/9.6 μg (PT003) | GFF MDI 1.2/9.6 μg (PT003) | FF MDI 9.6 μg (PT005) | Spiriva
Serious Adverse Events (participants affected / at risk) | 1/66 | 1/71 | 0/70 | 0/67 | 1/71 | 2/68 | 1/73 | 0/71
Other Adverse Events (participants affected / at risk) | 8/66 | 2/71 | 8/70 | 5/67 | 9/71 | 2/68 | 8/73 | 6/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI 18 μg (PT001) (N=66) | GFF MDI 18/9.6 μg (PT003) (N=71) | GFF MDI 9/9.6 μg (PT003) (N=70) | GFF MDI 4.6/9.6 μg (PT003) (N=67) | GFF MDI 2.4/9.6 μg (PT003) (N=71) | GFF MDI 1.2/9.6 μg (PT003) (N=68) | FF MDI 9.6 μg (PT005) (N=73) | Spiriva (N=71)
Cardio-Respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient Ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI 18 μg (PT001) (N=66) | GFF MDI 18/9.6 μg (PT003) (N=71) | GFF MDI 9/9.6 μg (PT003) (N=70) | GFF MDI 4.6/9.6 μg (PT003) (N=67) | GFF MDI 2.4/9.6 μg (PT003) (N=71) | GFF MDI 1.2/9.6 μg (PT003) (N=68) | FF MDI 9.6 μg (PT005) (N=73) | Spiriva (N=71)
Dry Mouth (Gastrointestinal disorders) | 8 (8) | 2 (2) | 3 (3) | 3 (3) | 5 (5) | 1 (1) | 6 (8) | 6 (6)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.